CLINICAL TRIAL: NCT04456270
Title: Asthma Control in a Dutch Primary Care Population
Status: Completed | Type: Observational
Sponsor: General Practitioners Research Institute (Network)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: GPRI19103
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Asthma; Asthma; Eosinophilic; Asthma Chronic; Asthma; Status
MeSH Terms: conditions — Asthma; Pulmonary Eosinophilia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary care patients with current asthma: Male and female primary care patients aged ≥18 years of age with clinically diagnosed asthma.

SUMMARY:
Rationale: Despite the availability of effective treatment to reach symptom control, nearly half of the asthma patients remain inadequately controlled. There is a need for timely and appropriate treatment of patients with uncontrolled asthma. Improving asthma control could be achieved by a better identification of causes followed by remediating modifiable factors in primary care or referral to secondary care. However, major gaps in evidence-based asthma practice exist in primary care. So far, there is a lack of knowledge on the prevalence of inadequate asthma and associated characteristics.

Objective: The primary objective is to determine the proportion of primary care patients with inadequate asthma control, as assessed during a regular control consultation with the general practice nurse.

Study design: This is a non-interventional prospective observational study, taking place in a real-world primary care setting. The AsthmaOptimiser tool will be used during regular asthma consultations in primary care, which the healthcare provider will fill in together with the patient. The AsthmaOptimiser tool creates an overview of factors and characteristics that may be associated with uncontrolled asthma, and subsequently provides a guideline-based management suggestion. Additionally, we will perform qualitative interviews to collect experiences and perspectives of healthcare providers on their use of the AsthmaOptimiser tool, including, but not limited to, ease of use, points of improvement, and on their implementation of the management suggestions.

Study population: Patients diagnosed with asthma, who attend a pre-planned primary care asthma review, are eligible to participate. A limited number of in- and exclusion criteria will be adopted, to make sure the research population closely resembles the real world.

Main study parameters/endpoints: The primary endpoint is the proportion of patients with inadequate asthma control. Inadequate asthma control will be defined as an exacerbation in the past 4 weeks and/or an ACQ6 (i.e., Asthma Control Questionnaire) score >0.75.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Physician diagnosis of Asthma
* Capacity to provide written informed consent

Exclusion Criteria:

* Life expectancy of less than 1 year
* Inability to understand Dutch
* Any other condition which, at the GPs and/or investigator's discretion, is believed to present a safety risk or may impact the study results
* Patients participating in a clinical trial that may distort outcomes in this observational study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Primary care patients with a current asthma diagnosis, who are scheduled to have in-person asthma review consultations with a primary care nurse, will be recruited from primary care practices located in the northern part of the Netherlands. The population includes men and women ≥18 years of age with clinically diagnosed asthma. The diagnosis of asthma is allowed to be a clinical diagnosis rendered by a doctor, without the requirement to conduct additional confirmatory testing. Furthermore, a limited number of in- and exclusion criteria will be adopted, to make sure the research population closely resembles the real world.
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Asthma Control Questionnaire | week prior to visit to general practice nurse for check-up appointment
  self-reported assessment of asthma symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Janwillem Kocks, PhD, Principal Investigator — General Practitioners Research Institute
Locations (1):
- GPRI, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided